CLINICAL TRIAL: NCT01902459
Title: A Non-Investigational Post-Market Trial Using EVARREST™ Fibrin Sealant Patch as an Adjunct to Hemostasis in Soft Tissue Bleeding During Intra-Abdominal, Retroperitoneal, Pelvic and Non-Cardiac Thoracic Surgery
Brief Title: EVARREST™ Fibrin Sealant Patch Post-Market Study
Acronym: EVARREST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 400-12-005
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Results first posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Hemorrhage; Soft Tissue Bleeding
Keywords: Hemostasis
MeSH Terms: conditions — Hemorrhage | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- EVARREST™ Fibrin Sealant Patch (Active Comparator): EVARREST™ Fibrin Sealant Patch consists of human fibrinogen and human thrombin embedded in a flexible composite patch component.
  Interventions: Biological: EVARREST™ Fibrin Sealant Patch
- Standard of Care (Other): Standard of Care (SoC) is manual compression with or without a topical absorbable hemostat.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Biological: EVARREST™ Fibrin Sealant Patch — EVARREST™ Fibrin Sealant Patch is a sterile, bio-absorbable combination product, comprised of two biological components (human plasma-derived fibrinogen and thrombin) embedded in a flexible composite patch component.
  Arms: EVARREST™ Fibrin Sealant Patch
Other: Standard of Care — Standard of Care will be manual compression (MC) with or without a topical absorbable hemostat (TAH) or any other adjunctive hemostasis technique that is deemed by the surgeon to be his/her standard of care.
  Arms: Standard of Care

SUMMARY:
The objective of this study is to evaluate the clinical utility of EVARREST™ Fibrin Sealant Patch (Fibrin Pad) as an adjunct to hemostasis in soft tissue bleeding during intra-abdominal (stomach area), retroperitoneal (hip and stomach area), pelvic (hip area) and non-cardiac thoracic (chest area) surgery.

DETAILED DESCRIPTION:
This is a randomized, controlled single-center study observing the clinical utility of EVARREST™ against standard of care (SoC) in controlling soft tissue bleeding. Standard of care will be manual compression (MC) with or without a topical absorbable hemostat (TAH) or any other adjunctive hemostasis technique that is deemed by the surgeon to be his/her standard of care. All subjects will be followed post-operatively through discharge and at 30 (+/-14) days.

Approximately 150 qualified subjects undergoing intra-abdominal, retroperitoneal, pelvic and non-cardiac thoracic surgery requiring adjunctive support for hemostasis for soft tissue bleeding will be enrolled in the study. Subjects will be randomized on a 1:1 basis, EVARREST™ vs. SoC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years of age, requiring an elective or urgent, open intra-abdominal, retroperitoneal, pelvic or non-cardiac thoracic surgical procedures;
* Subjects or legally authorized representative must be willing to participate in the study and provide written informed consent.
* Presence of an appropriate Target Bleeding Site as identified intra-operatively by the surgeon;

Exclusion Criteria:

* Subjects with known intolerance to blood products or to one of the components of EVARREST™ or unwilling to receive blood products;
* Female subjects who are pregnant or nursing.
* TBS is from a large defect in an artery or vein where the injured vascular wall requires repair and maintenance of vessel patency or where there would be persistent exposure of EVARREST™ to blood flow and/or pressure during absorption of the product;
* TBS with major arterial bleeding requiring suture or mechanical ligation;
* TBS within a contaminated or infected area of the body;
* Bleeding site is in, around, or in proximity to foramina in bone, or areas of bony confine;
* Subjects with any intra-operative findings identified by the surgeon that may preclude conduct of the study procedure;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2015-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kocharian, MD, Study Director — Ethicon, Inc.
Locations (1):
- Clinical Site #10, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Study endpoints

REFERENCES:
- [Derived] Ma GW, Kucey A, Tyagi SC, Papia G, Kucey DS, Varcoe RL, Forbes T, Neville R, Dueck AD, Kayssi A. The role of sealants for achieving anastomotic hemostasis in vascular surgery. Cochrane Database Syst Rev. 2024 May 2;5(5):CD013421. doi: 10.1002/14651858.CD013421.pub2. PMID 38695613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from July 2, 2013 through August 13, 2015 at a single center in the United States
Groups:
- EVARREST Fibrin Sealant Patch: EVARREST® Fibrin Sealant Patch is a sterile bio-absorbable combination product consisting of two constituent parts - a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin.
- Standard of Care (SoC): Manual compression with or without a topical absorbable hemostat
Period: Overall Study
Arm/Group | EVARREST Fibrin Sealant Patch | Standard of Care (SoC)
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat analysis set consisting of all randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | EVARREST Fibrin Sealant Patch | Standard of Care (SoC) | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Customized [Number; unit: Participants]
  18 to < 50 years | 23 | 20 | 43
  50 to < 65 years | 31 | 35 | 66
  65 to < 75 years | 15 | 16 | 31
  >= 75 yeatrs | 6 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 39 | 81
  Male | 33 | 36 | 69
Race/Ethnicity, Customized [Number; unit: Participants]
  White / Caucasian | 69 | 66 | 135
  Black or African American | 5 | 9 | 14
  Other | 1 | 0 | 1
BMI Category [Number; unit: Participants] — Underweight: < 18.5 kg/m^2, Normal weight: 18.5 - <25 kg/m^2, Overweight: 25 - <30 kg/m^2, Obese: 30 - <40 kg/m^2, Morbidly obese: 40 kg/m^2 or more
  Participants
    Underweight | 2 | 0 | 2
    Normal | 10 | 11 | 21
    Overweight | 15 | 22 | 37
    Obese | 37 | 34 | 71
    Morbidly obese | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Safety Parameter - Incidence of Thromboembolic Events
Description: Number of subjects experiencing a thromboembolic event as reported in the adverse events/serious adverse event safety set. the Safety set consists of all subjects on whom procedure is started.
Time Frame: Surgery up until the 30 day follow-up
Measure: Number; unit: Participants
Arm/Group | EVARREST Fibrin Sealant Patch | Standard of Care (SoC)
Number analyzed (Participants) | 75 | 75
Participants | 2 | 7

2. Primary Outcome: Safety Parameter - Incidence of Post-operative Bleeding Events Specifically Related to the Target Bleeding Site (TBS)
Description: Number of subjects experiencing a post-operative bleeding event specifically related to the target bleeding site (TBS) and as reported in the adverse events/serious adverse event safety set. Safety set consisting of all subjects on whom procedure is started.
Time Frame: Surgery up until the 30 day follow-up
Measure: Number; unit: Participants
Arm/Group | EVARREST Fibrin Sealant Patch | Standard of Care (SoC)
Number analyzed (Participants) | 75 | 75
Participants | 0 | 0

3. Primary Outcome: Safety Parameter - Incidence of Increase Blood Fibrinogen Level
Description: Number of subjects experiencing an increase in blood fibrinogen from the safety set consisting of all subjects on whom procedure is started.
Time Frame: Surgery up until the 30 day follow-up
Measure: Number; unit: Participants
Arm/Group | EVARREST Fibrin Sealant Patch | Standard of Care (SoC)
Number analyzed (Participants) | 75 | 75
Participants | 3 | 1

4. Other Pre Specified Outcome: This Product is Easy and Quick to Prepare for Application to the Target Bleeding Site.
Description: This product is easy and quick to prepare for application to the target bleeding site.
Time Frame: Intraoperative
Measure: Number; unit: Participants
Arm/Group | EVARREST Fibrin Sealant Patch | Standard of Care (SoC)
Number analyzed (Participants) | 75 | 75
Participants
  Strongly Disagree | 1 | 5
  Disagree | 0 | 0
  Neutral | 0 | 46
  Agree | 12 | 10
  Strongly Agree | 62 | 14

5. Other Pre Specified Outcome: This Product is Easy to Apply to a Variety of Bleeding Sites.
Description: This product is easy to apply to a variety of bleeding sites.
Time Frame: Intraoperative
Measure: Number; unit: Participants
Arm/Group | EVARREST Fibrin Sealant Patch | Standard of Care (SoC)
Number analyzed (Participants) | 75 | 75
Participants
  Strongly Disagree | 1 | 5
  Disagree | 0 | 1
  Neutral | 0 | 46
  Agree | 10 | 9
  Strongly Agree | 64 | 13
  Not applicable | 0 | 1

6. Other Pre Specified Outcome: This Product is Easy to Cut to Size for Application on Various Sized Bleeding Sites e.g., a Customized Preparation.
Description: This product is easy to cut to size for application on various sized bleeding sites e.g., a customized preparation.
Time Frame: Intraoperative
Measure: Number; unit: Participants
Arm/Group | EVARREST Fibrin Sealant Patch | Standard of Care (SoC)
Number analyzed (Participants) | 75 | 75
Participants
  Strongly Disagree | 1 | 5
  Disagree | 0 | 0
  Neutral | 0 | 45
  Agree | 7 | 8
  Strongly Agree | 66 | 15
  Not applicable | 1 | 2

ADVERSE EVENTS:
Time Frame: Surgical procedure through 30 (+/- 24 days) post surgery
Arm/Group | EVARREST Fibrin Sealant Patch | Standard of Care (SoC)
Serious Adverse Events (participants affected / at risk) | 3/75 | 7/75
Other Adverse Events (participants affected / at risk) | 6/75 | 10/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EVARREST Fibrin Sealant Patch (N=75) | Standard of Care (SoC) (N=75)
Deep vein thrombosis (Vascular disorders) | 0 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EVARREST Fibrin Sealant Patch (N=75) | Standard of Care (SoC) (N=75)
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less